CLINICAL TRIAL: NCT04438915
Title: The Effect of Obesity on the Incidence of Postoperative Cognitive Dysfunction in Gynecological Day-case Surgery
Brief Title: The Effect of Obesity on the Incidence of Postoperative Cognitive Dysfunction in Gynecological Day Case Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Hussein Bahr, Lecturer in Anaesthesia , Surgical ICU and Pain management department . Faculty of medicine ., Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FMBSUREC/03052020/Bahr
Record Dates: First submitted 2020-06-06; First posted 2020-06-19 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Obesity; Day-case Surgery; Postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications; Obesity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The doctor who ask the MMS is not informed about the design of the study .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Average weight .control group (No Intervention): Average weight BMI (18.5_25)
- Overweight (Active Comparator): Overweight BMI ( 25_30 )
  Interventions: Behavioral: Effect of Obesity on incidence of Postoperative cognitive in Gynecological Day- Day- case surgery
- Mild obese (Active Comparator): Mild obese BMI (30_35 )
  Interventions: Behavioral: Effect of Obesity on incidence of Postoperative cognitive in Gynecological Day- Day- case surgery

INTERVENTIONS:
Behavioral: Effect of Obesity on incidence of Postoperative cognitive in Gynecological Day- Day- case surgery — The effect of obesity on the incidence of postoperative cognitive dysfunction in Gynecological day-case surgery
  Arms: Mild obese; Overweight

SUMMARY:
Cognitive dysfunction is the impairment of mental process of perception. memory and information processing which allow the human to acquire knowledge and plan for the future. The etiology of Post operative cognitive dysfunction (POCD) is unclear and seems to be multifactorial involving a combination of patient, surgical, anesthetic and environmental factors. The definition of day surgery in Great Britain and Ireland is clear; the patient is admitted and discharged on the same day.

DETAILED DESCRIPTION:
Cognitive dysfunction is the impairment of mental process of perception. memory and information processing which allow the human to acquire knowledge and plan for the future. The etiology of Post operative cognitive dysfunction (POCD) is unclear and seems to be multifactorial involving a combination of patient, surgical, anesthetic and environmental factors. It can be a manifestation of transient or permanent cerebral injury. While cognitive function tends to improve overmonths to years postoperatively in affected individuals, some proportion has seemingly permanent cognitive injury. Most of the studies of POCD, however, have methodological difficulties, as pointed out by Newman and colleagues in their review of more than 40 studies.

The overweight/obese population has been steadily increasing worldwide. According to the WHO, with1.3 billion overweight (25 < body mass index [BMI] < 30) people and 600 million obese (BMI > 30) people in the world, the obesity rate exceeds10% for both genders and has more than doubled during the past 40 years. Furthermore, It considered as seven of the top10 causes of death / physical disability and chronic disorders such as cancer and diabetes, which are closely related to obesity.

The definition of day surgery in Great Britain and Ireland is clear; the patient is admitted and discharged on the same day, with day surgery as the intended management. The term '23-h stay' is used in the United states healthcare system. Obesity itself is not a contraindication to day surgery, as morbidly obese patients can be safely managed by experts, provided appropriate resources are available. This includes factoring in additional time for anaesthesia and surgery as well as the presence of skilled assistants and equipment.

The incidence of complications during the operation or in the early recovery phase is greater in patients with increasing body mass index. However, these problems would still occur with inpatient care and have usually resolved or been successfully treated by the time a day-case patient would be discharged. In addition, obese patients benefit from short-duration anaesthetic techniques and early mobilisation associated with day surgery.

Our study will aim to assess the early cognitive dysfunction after general anesthesia in normal weight patients, overweight and mild obese patients in gynacological day-case surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging 20_40 years, ASA physical status I undergoing hysteroscopy procedures
* All patients can read and write well

Exclusion Criteria:

Patients not ASA1 Patients receiving sedatives as midazolam. Pregnant Patients . Patients with cerebrovascular diseases . Patients with history of allergy to the drugs used in the study or patients with substance abuse .

Time of anesthesia less than 30 minute ,or more than one hour . Irrigation fluid rather than warm saline(40 degree ) or fluid volume more than 1500 ml

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gynecological Day- case surgery
Enrollment: 138 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction( POCD ) | 1 hour Preoperative _ then 1 hour , 6 hours and 24 hour postoperatively
  Mini Mental State a practical method for grading the cognitive state ( Max score 30 degree ) Orientation 10 degree , Registration 3 degree , Attention&Calculation 5 degree , Recall 3 degree , language 9 degree .
  Decrease 2 or more than Preoperative score will indicate POCD.

SECONDARY OUTCOMES:
weight ln kilograms (KG ) and Height in meters (M ) will be combined to report Body mass index (BMI ) . BMI = KG/ M^2 . | Preoperative.
  To show the effect of obesity on POCD
Vital signs: HR (beat/min), MAP (mmHg) and peripheral Oxygen saturation (Spo2) % | immediately prior to induction of anesthesia and subsequently every 5 min till the termination of anesthesia.
  To make other factors irrelevant
Time of surgery in minutes | Intraoperative
  To make other factors irrelevant
AGE in years | Preoperative
  To make other factors irrelevant

CONTACTS AND LOCATIONS:
Overall Officials: Amira F Elgaml, Study Director — Faculty of medicine.Beni-suef university
Locations (1):
- Faculty of medicine.Beni-suef university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The effect of obesity on the incidence of postoperative cognitive dysfunction in Gynecological Day- case surgery
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: The effect of obesity on the incidence of postoperative cognitive dysfunction in Gynecological Day- case surgery
URL: http://www.bsu.edu.eg